CLINICAL TRIAL: NCT02533583
Title: Pulse Oximetry With Clinical Observation to Screen for Lung Disease in Neonates
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, yangjie, professor, Guangdong Women and Children Hospital
Other Study IDs: guangdongwchhi1
Record Dates: First submitted 2015-08-04; First posted 2015-08-27 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Lung Diseases
Keywords: pulse oximetry; clinical assessment; neonate; lung disease
MeSH Terms: conditions — Lung Diseases | interventions — Oximetry

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- symptomatic newborn: the symptomatic newborn cohort( symptomatic definition see detail),all of babies will referred for chest X-ray,and within 2 hours performing echocardiography to exclude critical and serious heart disease.All clinical assessment will do by attending doctor.
  Interventions: Device: pulse oximetry (PHILIPS intelliven MP5)
- Asymptomatic newborn: the asymptomatic newborn cohort will gave pulse oximetry and clinical assessment every 8 hours within 3 days.everybody have positive results will been preformed chest X-ray and echocardiography.All clinical assessment will do by attending doctor.
  Interventions: Device: pulse oximetry (PHILIPS intelliven MP5)

INTERVENTIONS:
Device: pulse oximetry (PHILIPS intelliven MP5) — all newborn monitor pulse oximetry in left hand
  Other Names: PHILIPS intelliven MP5

SUMMARY:
The investigator assessed the feasibility and reliability of pulse oximetry plus clinical observation for detection the lung disease in neonates.

DETAILED DESCRIPTION:
At present respiratory disease(RDS) diagnose base on clinical symptom and chest X-ray.But in china, because of the difference of medical conditions, some areas especially the basic level hospitals without the condition of X-ray examination, which can not be clearly diagnosed RDS.In 2013, the scholars analyzed the disease of neonatal intensive care unit (NICU) need to be exposed to radiation, and RDS was in the first place. There is no conclusion whether it bad for newborn to exposure more. But in animal models, there is a correlation between exposure to radiation and cancer.

Hyaline membrane disease(HMD) is common occur in preterm infants .pulmonary surfactant(PS) is a safe and effective treatment for neonatalHMD.Bahadue F L meta analyse conclusion is early application of PS is more benefit for HMD.

So investigator hypothesize that pulse oximetry with clinical assessment have high sensitivity,specificity ,positive and negative predictive value to lung disease.The aim is to reduce radiation exposure to neonate and to preterm infants with RDS can early application of PS.

Symptomatic definition:with grunting,nasal flaring,retraction,cyanosis,tachypnea,stridor.

Pulse oximetry positive criteria:1.atrial oxygen saturation (SpO2)<90%;2.heart rate>180 or <100 per minute.

Clinical assessment:1.respiratory physical examination:non-symmetry,decrease breathing sound,bubbles sound.2.Delivery history:caesarean,premature rupture of membranes,liquor,mother conditions,Apgar score.

Congenital heart disease classification:1.critical:defects causing of the death or needing intervention before 28 days.2.serious:defects needing intervention before 1 year of age.significant:defects persisting longer than 6 months of age ,but not classified as critical or serious.4.non-significant:defects not physically appreciable and not persisting after 6 months of age.

ELIGIBILITY:
Inclusion Criteria:

1. gestation age :28 to 42 weeks
2. birth weight :1000-4000g
3. asymptomatic or symptomatic respiratory symptom

Exclusion Criteria:

1. gestation age <28 weeks or >42 weeks
2. birth weight <1000g or >4000g
3. critical and serious heart disease
4. congenital malformation

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants will born in guangdong women and children hospital
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
pulse oximetry with clinical observation screen lung disease sensitivity | 7 days
  use wilson method to calculate the sensitivity

SECONDARY OUTCOMES:
pulse oximetry with clinical observation screen lung disease specificity | 7 days
  use wilson method to calculate the specificity
pulse oximetry with clinical observation screen lung disease positive and negative value | 7 days
  use logistic regression model wo calculate the accuracy of the method

CONTACTS AND LOCATIONS:
Overall Officials: jie yang, doctor, Study Chair — Guangdong Women and Children Hospital

REFERENCES:
- [Background] Zhao QM, Ma XJ, Ge XL, Liu F, Yan WL, Wu L, Ye M, Liang XC, Zhang J, Gao Y, Jia B, Huang GY; Neonatal Congenital Heart Disease screening group. Pulse oximetry with clinical assessment to screen for congenital heart disease in neonates in China: a prospective study. Lancet. 2014 Aug 30;384(9945):747-54. doi: 10.1016/S0140-6736(14)60198-7. Epub 2014 Apr 22. PMID 24768155
- [Background] Iyer NP, Baumann A, Rzeszotarski MS, Ferguson RD, Mhanna MJ. Radiation exposure in extremely low birth weight infants during their neonatal intensive care unit stay. World J Pediatr. 2013 May;9(2):175-8. doi: 10.1007/s12519-013-0417-1. Epub 2013 May 16. PMID 23677834
- [Background] Bahadue FL, Soll R. Early versus delayed selective surfactant treatment for neonatal respiratory distress syndrome. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD001456. doi: 10.1002/14651858.CD001456.pub2. PMID 23152207